CLINICAL TRIAL: NCT06897371
Title: Effect of Postpartum Hemorrhage Management Education Given With Kahoot Method on Knowledge, Self-Confidence in Intervention and Motivation Levels of Midwifery Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBU-AYDINKARTAL-013
Record Dates: First submitted 2024-12-07; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Game-based Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (n:40) (Experimental): A 5-question trial test on Kahoot usage will be applied to the students in the intervention group (questions must be prepared in advance, students must have full internet connection, students must enter the Kahoot application with their phones, students must enter the code required to enter the platform, etc.). The questions that make up the trial test will be created independently of the subject covered in the theoretical training and students will be adapted to Kahoot. After the 2-hour theoretical training is completed, reinforcement will be provided using the 25-question game-based learning method on the Kahoot platform. Brief explanations will be made to reinforce the subject and the reinforcement session will last for 30 minutes. The "Self-Confidence/Competence Scale in Patient Intervention", "Postpartum Hemorrhage Management Information Form" and "Motivation Scale Regarding the Teaching Material" will be applied to both groups as a post-test.
  Interventions: Other: Games-based education
- Control group (n:40 (No Intervention): A 2-hour training will be given with a power point presentation, including theoretical information, case discussion and video demonstration on the evaluation and management of postpartum hemorrhage.

INTERVENTIONS:
Other: Games-based education — A 5-question trial test on Kahoot usage will be applied to the students in the intervention group (questions must be prepared in advance, students must have full internet connection, students must enter the Kahoot application with their phones, students must enter the code required to enter the platform, etc.). The questions that make up the trial test will be created independently of the subject covered in the theoretical training and students will be adapted to Kahoot. After the 2-hour theoretical training is completed, reinforcement will be provided using the 25-question game-based learning method on the Kahoot platform. Brief explanations will be made to reinforce the subject and the reinforcement session will last for 30 minutes. The "Self-Confidence/Competence Scale in Patient Intervention", "Postpartum Hemorrhage Management Information Form" and "Motivation Scale Regarding the Teaching Material" will be applied to both groups as a post-test.
  Arms: Intervention group (n:40)

SUMMARY:
This study was planned to investigate the effect of postpartum hemorrhage management training given with the Kahoot method on the knowledge, self-confidence in intervention and motivation levels of midwifery students. The research population will consist of third-year students studying at the Department of Midwifery, Hamidiye Faculty of Health Sciences (HSBF), Health Sciences University (SBU) in the spring semester of the 2024-2025 academic year (N: 80). In this semi-experimental pre-test and post-test design and control group planned study, in order to determine the sample size; the data were normally distributed, the standard deviation of the main mass was estimated as 1 and the effect size (effect size, difference) was estimated as 0.8. For the analysis to be conducted, it was calculated that the highest power value of the study would be 0.942182 if two independent n₁=40, n₂=40 samples were taken at a significance level of 5%. In addition, the adequacy of the sample size in the study will be evaluated with post hoc power analysis after the data are collected.

Students who volunteer to participate in the study will be assigned to the intervention and control groups using the computer-aided simple random sampling method. Computer-aided randomization will be used in the study, and the number of cases will be entered through the program with the URL address https://www.randomizer.org and random assignment will be made to the intervention and control groups. Before the data collection forms begin training, the "Informed Voluntary Consent Form" will be shared with the students participating in the study and their approval will be requested. The "Introductory Information Form", "Postpartum Hemorrhage Management Information Form", "Self-Confidence/Competence Scale in Patient Intervention" and "Motivation Scale Regarding the Teaching Material" will be applied to the students who agree to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research.
* Having internet access,
* Having a smart phone,
* Being an active student in the 3rd year of the Department of Midwifery at Hamidiye Health Sciences Faculty, University of Health Sciences.

Exclusion Criteria:

* Being a passive student in the 3rd year of the Midwifery Department of Hamidiye Health Sciences Faculty, University of Health Sciences.
* Not meeting the inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2025-11-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 10 minutes
  This form, created by researchers based on literature, includes questions about the participants' age, high school graduation, whether they choose the profession willingly, whether they feel they belong to the profession, et
Postpartum Hemorrhage Management Information Form | 10 minutes
  The form was created by researchers based on literature and structured as multiple choice and true-false, and finalized with expert opinion (16, 17, 18). 25 multiple choice (12 questions) and true-false (13 questions) questions were prepared, which were considered appropriate for the purpose of the study and the educational content. The form's success evaluation will be carried out out of 100 points. For this purpose, the students' total success points were calculated as 4 times the number of correct answers. Students will be evaluated by giving "4" points for each correct answer and "0" points for each wrong answer. The highest score that students can get from the information form was determined as "100" and the lowest score was determined as "0".
Self-Confidence/Competence in Patient Intervention Scale | 10 minutes
  The validity and reliability study of the scale was conducted by Terzioğlu et al. in 2012. In the explanatory factor analysis of the scale developed for health professional students, 3 factors were obtained. The three factors were classified as clinical practice (11 items), psychological support (4 items), and health care system knowledge (3 items). The validity results of the scale were evaluated between 0.80 and 0.94. The Cronbach Alpha internal consistency coefficient of the scale is 0.947. The scale contains a total of 18 items and is evaluated according to the 5-point Likert system (1=Strongly Disagree, 2=Disagree, 3=Undecided, 4=Agree, 5=Strongly Agree). The highest score that can be obtained from the scale was determined as 55, and the lowest score was determined as 11.
Motivation Scale Related to Instructional Material | 10 minutes
  The scale was developed by Keller, who evaluated the entire course, in order to measure motivations related to the instructional material, based on the ARCS (Attention, Relevance, Confidence, Satisfaction) Model (20). The Turkish adaptation of the scale was carried out by Dinçer and Doğanay. The scale, designed with a five-point Likert type (Very True=5, True=4, Moderately True=3, Somewhat True=2, Not True=1), consists of 33 items and four sub-dimensions (attention, suitability, confidence, satisfaction). The highest score that can be obtained from the attention dimension is 50, the lowest score is 10. The highest score that can be obtained from the suitability dimension is 40, the lowest score is 8. The highest score that can be obtained from the confidence dimension is 45, the lowest score is 9.

SECONDARY OUTCOMES:
Introductory Information Form | 10 minutes
  This form, created by researchers based on literature, includes questions about the participants' age, high school graduation, whether they choose the profession willingly, whether they feel they belong to the profession, et
Postpartum Hemorrhage Management Information Form | 10 minutes
  The form was created by researchers based on literature and structured as multiple choice and true-false, and finalized with expert opinion (16, 17, 18). 25 multiple choice (12 questions) and true-false (13 questions) questions were prepared, which were considered appropriate for the purpose of the study and the educational content. The form's success evaluation will be carried out out of 100 points. For this purpose, the students' total success points were calculated as 4 times the number of correct answers. Students will be evaluated by giving "4" points for each correct answer and "0" points for each wrong answer. The highest score that students can get from the information form was determined as "100" and the lowest score was determined as "0".
Self-Confidence/Competence in Patient Intervention Scale | 10 minutes
  The validity and reliability study of the scale was conducted by Terzioğlu et al. in 2012. In the explanatory factor analysis of the scale developed for health professional students, 3 factors were obtained. The three factors were classified as clinical practice (11 items), psychological support (4 items), and health care system knowledge (3 items). The validity results of the scale were evaluated between 0.80 and 0.94. The Cronbach Alpha internal consistency coefficient of the scale is 0.947. The scale contains a total of 18 items and is evaluated according to the 5-point Likert system (1=Strongly Disagree, 2=Disagree, 3=Undecided, 4=Agree, 5=Strongly Agree). The highest score that can be obtained from the scale was determined as 55, and the lowest score was determined as 11.
Motivation Scale Related to Instructional Material | 10 minutes
  The scale was developed by Keller, who evaluated the entire course, in order to measure motivations related to the instructional material, based on the ARCS (Attention, Relevance, Confidence, Satisfaction) Model (20). The Turkish adaptation of the scale was carried out by Dinçer and Doğanay. The scale, designed with a five-point Likert type (Very True=5, True=4, Moderately True=3, Somewhat True=2, Not True=1), consists of 33 items and four sub-dimensions (attention, suitability, confidence, satisfaction). The highest score that can be obtained from the attention dimension is 50, the lowest score is 10. The highest score that can be obtained from the suitability dimension is 40, the lowest score is 8. The highest score that can be obtained from the confidence dimension is 45, the lowest score is 9.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No